CLINICAL TRIAL: NCT05920447
Title: Safety and Limitation of the 2nd Generation Laryngeal Mask Airway in the Lithotomy Position: An Obsevational Study
Acronym: LMA
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU R 76/2021
Record Dates: First submitted 2023-05-26; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-05

CONDITIONS: Airway Management

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ETT: the patients in group T were intubated with Endotracheal tube (ETT) (flexicare) size 7 for female and 8 for male
  The patients were ventilated with a volume-controlled mode at a Tidal Volume (TV) 7ml/kg, Respiratory Rate 12 /min, I: E 1:2. The patient was then positioned in the lithotomy position.
  Ventilatory parameters including expired TV, peak airway pressure, inspired- expired TV and the end-tidal carbon dioxide were all monitored and recorded every 5 min.
  In case of leaking from the LMA that interfere with the ventilation before the patients were being positioned in the lithotomy position, the patients were excluded and replaced by another.
  The incidence of aspiration as revealed clinically( witnessed vomiting followed by decreased oxygen saturation, increased airway pressure, tachycardia, etc..) and confirmed radiologically, Failure of insertion or intubation, sore throat and air leak were reported as a complications.
- LMA: The patients in group L were intubated with an I gel Laryngeal mask airway (LMA) , the size was selected based on the body weight according to the manufacturer's instructions,
  The patients were then ventilated with a volume-controlled mode of ventilation at a Tidal Volume (TV) 7ml/kg, Respiratory Rate 12 /min, I: E 1:2. The patient was then positioned in the lithotomy position and secured
  Ventilatory parameters including expired TV, peak airway pressure, TV inspired- TV expired and the end-tidal CO2 were all monitored and recorded every 5 min.
  In case of leaking from the LMA that interfere with the ventilation before the patients were being positioned in the lithotomy position.
  The incidence of aspiration as revealed clinically( witnessed vomiting followed by decreased oxygen saturation, increased airway pressure, tachycardia, etc..) and confirmed radiologically, Failure of insertion or intubation, sore throat and air leak were reported as a complications.
  Interventions: Device: LMA

INTERVENTIONS:
Device: LMA — Monitor the ventilatory parameter and incidence of complications
  Groups: LMA

SUMMARY:
Laryngeal mask airway is used in different types of surgery requiring different position, recommendation was raised regarding the use of LMA in Lithotomy position with pressure controlled mode of ventilation. This raise a concern whether the mode of ventilation is a limitation for the use of LMA in these position, especially with the use of the i-gel LMA with the characteristic non-inflatable jelly cuff, that provides an excellent seal.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Both gender
* Surgery mandating lithotomy position

Exclusion Criteria:

* Patients' refusal
* Pregnant women
* Obesity (BMI > 39)
* Trendelenburg position
* Moderate to severe GERD
* Lengthy procedures (more than 120 min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients in group L were intubated with an Igel LMA (Intersurgical) , the size was selected based on the body weight according to the manufacturer's instructions, the patients in group T were intubated with ETT (flexicare) size 7 for female and 8 for male
  The patients were then ventilated with a volume-controlled mode of ventilation at a Tidal Volume (TV) 7ml/kg, Respiratory Rate 12 /min, I: E 1:2. The patient was then positioned in the lithotomy position and secured
  Ventilatory parameters including expired TV, peak airway pressure, TV inspired- TV expired and the end-tidal CO2 were all monitored and recorded every 5 min.
  The incidence of aspiration as revealed clinically( witnessed vomiting followed by decreased oxygen saturation, increased airway pressure, tachycardia, etc..) and confirmed radiologically, Failure of insertion or intubation, sore throat and air leak were reported as a complications.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-24 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Assess the safety of volume-controlled mode of ventilation.in the Lithotomy position during the procedure | During the Procedure
  Measuring the air Leak through measuring the difference between the inspired and expired tidal volume and determine the peak airway pressure at which these leak does occur.

SECONDARY OUTCOMES:
THE incidence of complication among the two groups | through the procedure
  decreased oxygen saturation, increased airway pressure, tachycardia, etc..) and confirmed radiologically, Failure of insertion or intubation, sore throat and air leak were reported as a complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No